CLINICAL TRIAL: NCT02015949
Title: The Control of Brain Networks After Traumatic Brain Injury: a Neuroimaging and Neuropsychological Study of Dopamine and Cognition
Brief Title: The Relationship Between Traumatic Brain Injury and Dopamine (a Chemical in the Brain)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13HH1824; 2013-004244-37 (EudraCT Number)
Record Dates: First submitted 2013-11-25; First posted 2013-12-19 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Active Comparator): 2 weeks of 0.3mg/kg twice daily of methylphenidate to the nearest 5mg
  Interventions: Drug: Methylphenidate
- Sugar pill (Placebo Comparator): 2 weeks of twice daily placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Cross-over design comparing methylphenidate 0.3 mg/kg (to nearest 5mg) twice daily to placebo
  Arms: Methylphenidate
Drug: Placebo — Twice daily placebo tablet for two weeks
  Arms: Sugar pill

SUMMARY:
Traumatic brain injury (TBI) is the most common cause of death and disability in young adults. Patients can experience significant problems with concentration, attention, and memory (so called 'cognitive impairments') following TBI. These cognitive impairments can drastically impact on a patient's well-being, and can lead to significant economic and social consequences. Roughly a quarter of TBI patients improve but an equal number deteriorate over time. The investigators know little about why patients vary so much in how they recover. Crucially, the investigators have no treatments to improve brain functioning or recovery after TBI.

Trials investigating ways of protecting the brain just after injury have been disappointing. An alternative strategy, however, is to improve the function of brain regions that remain intact, but that function inefficiently after TBI. The investigators know that dopamine (a chemical in the brain) is known to influence many brain functions and the investigators know that pathways in the brain that use dopamine are affected by TBI.

In humans, drugs that increase dopamine in the brain, such as methylphenidate, are sometimes used to enhance cognitive function after TBI, but the response to treatment can be highly variable between patients. Therefore, what is needed in the clinic is a way to target the use of these drugs to patients who are likely to respond.

In a single centre study, the investigators will use SPECT (Single Photon Emission Tomography) imaging to measure dopamine levels in the brain. MRI (Magnetic Resonance Imaging) scans will assess brain structure and function. The investigators will test whether treatment with methylphenidate improves cognitive functions in TBI patients who have ongoing cognitive problems, whether the mechanism involves a normalisation of brain functioning and whether brain dopamine levels can predict the magnitude of any improvement in symptoms.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of a moderate-severe traumatic brain injury (as defined by the Mayo TBI severity classification system) at least 3 months prior to recruitment into the study
* age between 20 and 65 years
* capable of giving written informed consent subjective complaint of cognitive difficulties by the participant, treating clinician, or caregiver

Exclusion Criteria:

* unwillingness or inability to follow the procedures required
* significant neurological or psychiatric illness diagnosed prior to the TBI
* family history of a first degree relative with a psychotic illness
* currently participating in a clinical trial or has done so within 1 month before screening
* use of any medication or substance that, in the opinion of the investigators, would interfere with the study or compromise participant safety
* history of a drug or other allergy that, in the opinion of the investigators, contraindicates their participation in the study
* history of current or past drug or alcohol addiction
* female participants who are breast feeding or pregnant (positive pregnancy test) or plan to become pregnant during the study
* positive urine drug screen
* contraindication to MRI scanning, assessed by a standard pre-MRI questionnaire
* contraindication to the use of methylphenidate (including medications deemed to have a potentially serious interaction with methylphenidate as per the British National Formulary)
* clinical evidence of motor symptoms of Parkinsonism as assessed by a Neurologist

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The change in Choice Reaction Time task with methylphenidate treatment in patients and its relationship to specific binding ratio (SBR) of the dopamine transporter (DAT) in the striatum. | On completion of the four week drug trial phase

CONTACTS AND LOCATIONS:
Overall Officials: David J Sharp, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, London, United Kingdom